CLINICAL TRIAL: NCT00512720
Title: Clinical Outcomes of Three Different Percutaneous Revascularization Strategies for the Treatment of Lifestyle Limiting Claudication: A Retrospective Analysis
Acronym: FIX-IT Retro
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: West Michigan Heart (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2007-174
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Artery Disease
Keywords: PAD; Peripheral Artery Disease; PVD; Peripheral Vascular Disease; Leg Blockage; Angioplasty; Stent; Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Intermittent Claudication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine the effect of three different percutaneous revascularization strategies (Balloon Cryoplasty vs. Stent Placement vs. Atherectomy) in the treatment of lifestyle limiting lower extremity claudication

DETAILED DESCRIPTION:
Endovascular revascularization of the superficial femoral artery (SFA) has become one of the most commonly performed endovascular procedures.The ability to offer the patient an alternative to surgical revascularization, limited by significant morbidity and mortality, with a same-day outpatient percutaneous procedure underlies the popularity of the endovascular approach. Although surgical bypass of the SFA remains the gold standard for revascularization, it is associated with significant morbidity and mortality.Comparative data between cryoplasty, angioplasty or stenting of the SFA will ultimately be required to provide more robust evidence of the efficacy of each mode of therapy.This registry is designed to determine the efficacy of three different percutaneous revascularization strategies (Cryoplasty vs. Stent Placement vs. Atherectomy) in the treatment of lifestyle limiting lower extremity claudication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Superficial Femoral Artery disease as assessed by angiography

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female over the age of 18 who have had Three Different Percutaneous Revascularization Strategies
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2007-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mustapha, MD, Principal Investigator — Corewell Health West; Dennis Dunning, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States